CLINICAL TRIAL: NCT02381730
Title: Assessment of Visual Acuity in Patients With Polypoidal Choroidal Vasculopathy and Aflibercept Treatment
Acronym: PCV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-A01717-38
Record Dates: First submitted 2015-03-05; First posted 2015-03-06 (Estimated); Last update posted 2017-12-08 (Actual); Status verified 2017-12

CONDITIONS: Polypoidal Choroidal Vasculopathy
MeSH Terms: conditions — Polypoidal Choroidal Vasculopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Aflibercept (Experimental)
  Interventions: Drug: Intravitreal aflibercept

INTERVENTIONS:
Drug: Intravitreal aflibercept — Patient receive one intravitreal injection of 2mg aflibercept (as currently recommended in the treatment of AMD)

SUMMARY:
Polypoidal choroidal vasculopathy (PCV) is a disease of the choroidal vasculature, that is often regarded as a sub-type of age-related macular degeneration (AMD). However, PCV response to anti-vascular agents differs from the response of typical AMD.

This study aims at describing the evolution of the best corrected visual acuity (BCVA) in PCV patients, 28 weeks after they receive one injection of intravitreal aflibercept (2mg).

ELIGIBILITY:
Inclusion Criteria:

* Active polypoidal choroidal vasculopathy,
* Visual acuity superior to 1/10 (20/200) and inferior to 6,25/10 (20/32)
* Age above 45
* No prior intravitreal treatment, or no response to prior treatment by 3 injections of ranibizumab, or disease recurrence after more than 3 months of stability
* Intravitreal injection of aflibercept is indicated by current clinical recommendations

Exclusion Criteria:

* Simultaneous treatment with another anti-VEGM agent
* Diabetic retinopathy
* Personal history of vitrectomy or uveitis
* Personal history laser photocoagulation and/or verteporphin phototherapy
* Tear in the pigmentary epithelium
* Chorioretinitis scar
* Macular atrophy in the pigmentary epithelium
* Treatment with corticosteroids
* Eye surgery less than 3 months before inclusion

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2014-01; Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Evolution of the best corrected visual acuity (BCVA) measured on the EDTRS scale, between pre-injection and 28 weeks after injection | 28 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Martine Mauget-Faysse, Principal Investigator — Fondation Ophtalmologique A. de Rothschild
Locations (3):
- France (3):
  - CHU Lyon Croix Rousse, Lyon
  - Fondation Ophtalmologique A. de Rothschild, Paris
  - Centre Médical de la Rétine Maison Rouge, Strasbourg